CLINICAL TRIAL: NCT04834531
Title: Effect of Zhuli Capsule on Phlegm-heat Syndrome (Tan-re Zheng) in the Acute Exacerbations of Chronic Obstructive Pulmonary Disease or Chronic Bronchitis
Brief Title: Effect of Zhuli Capsule on Phlegm-heat Syndrome (Tan-re Zheng)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Institute of Clinical Basic Medicine of Traditional Chinese Medicine, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZLJN-V2.0
Record Dates: First submitted 2020-09-21; First posted 2021-04-08 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zhuli capsule (Experimental): Base on the standard medical treatment, the patients in this group will be used Zhuli capsule, 2 capsules (1.2 g) once, three time a day for 7 days.
  Interventions: Drug: Zhuli capsule; Other: Standard medical treatment
- Placebo (Placebo Comparator): Base on the standard medical treatment, the patients in this group will be used placebo capsule, 2 capsules (1.2 g) once, three time a day for 7 days.
  Interventions: Drug: Placebo; Other: Standard medical treatment

INTERVENTIONS:
Drug: Zhuli capsule — This capsule is made from the exact of Phyllostachys glauca McClure or Phyllostachysnuda McClure, which has the expectorant effects. It is oral used,2 capsules for once, three times a day, for 7 days.
  Arms: Zhuli capsule
Drug: Placebo — The placebo capsule is filled with amylodextrin made with food colour and flavor，with the similar appearance, smell and flavor with Zhuli Capsule. It is oral used, 2 capsules for once, three times a day, for 7 days.
  Arms: Placebo
Other: Standard medical treatment — Standard medical treatment will be given according to the recent guidelines with the evaluation of the clinicians, include:
  1. if the patient with AECOPD, he or she will be given with oxygen therapy, bronchodilators, glucocorticoid or antibacterial drugs;
  2. if the patient with AECB, he or she will be given with antibacterial drugs or anti-asthmatic drugs for asthma attacks.

SUMMARY:
This trial aims to evaluate the clinical control rate of sputum by Zhuli Capsule in the treatment of the Phlegm-heat Syndrome （Tan-re Zheng）in the patients with acute exacerbation of chronic obstructive pulmonary disease or chronic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of acute exacerbation in chronic obstructive pulmonary disease or chronic bronchitis;
2. Meet the diagnostic criteria of Phlegm-heat Syndrome (Tan-re Zheng) in TCM
3. Age from 18 to 75 years old, regardless of gender;
4. The score of each dimension of the sputum assement scale is ≥1;
5. Those who have not participated in other drug clinical research in the past one month;
6. Sign the informed consent letter.

Exclusion Criteria:

1. Patients with pulmonary tuberculosis, bronchial cancer or other lung diseases.
2. Loose stools due to Spleen deficiency and stomachache caused by cold.
3. Diabetes or severe cardiovascular, liver (ALT>1.5×ULN), kidney (Cr>1.5×ULN) and other primary diseases.
4. Pregnant and lactating women.
5. Patients with acute and chronic respiratory failure.
6. Those who cannot give full informed consent due to mental disorders.
7. People with disabilities recognized by law.
8. People with allergies, or allergic to the ingredients of the drug used in this test.
9. Those who have used drugs with expectorant effects within the day.
10. Patients who are participating in clinical trials of other drugs. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The clinical control rate of sputum | Day 7
  Defined as the proportion of patients with the expectoration rate ≥90%.

SECONDARY OUTCOMES:
Time to sputum turn white | up to Day 7
Cough Symptom Score Scale | 0,Day 3, Day 7
  Cough Symptom Score Scale include Day Cough Symptom Score and Night cough symptom score. In Day Cough Symptom Score, zero means no cough,one means occasionally short cough,two means frequent cough, slightly affecting daily activities,three means frequent coughing seriously affects daily activities;In Night cough symptom score,zero means no cough,one means short-term cough when falling asleep or occasional night cough,two means cough slightly affects night sleep,three means cough seriously affects night sleep.
Use of Antibiotic | 0,Day 3, Day 7
Chronic obstructive pulmonary disease Assessment Test | 0,Day 3, Day 7
The Phlegm-heat Syndrome (Tan-re Zheng) scale | 0,Day 3, Day 7
  The Phlegm-heat Syndrome (Tan-re Zheng) scale include measures of the main symptoms and the secondary symptoms. The main symptom is about the color ，the characteristics and the amount of sputum.Each one includes four levels,0 represents normal，3 represents mild symptom,6 represents moderate symptom,9 represents Severe symptom.The secondary symptoms include Day cough，Night cough，Dry throat thirst，fever，blush，Dry stool，Yellow urine ，Red tongue and pulse.Each one includes different levels.The higher score represents the more meeting The Phlegm-heat Syndrome (Tan-re Zheng) ，the lower score means the opposite.
The change value about the volume of sputum after treatment | 0,Day 3, Day 7
  Monitor the sputum volume everyday and compare changes in sputum volume in the treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Sichuan Provincial Hospital of Traditional Chinese Medicine, Chengdu, Sichuan
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou, Zhejiang